CLINICAL TRIAL: NCT03781466
Title: Effect of Cervical Cerclage With or Without Vaginal Progesterone Versus Vaginal Progesterone Alone for Prevention of Preterm Labor in Asymptomatic Twin Pregnancies With a Sonographic Short Cervix: A Randomized Clinical Trial
Brief Title: Effect of Cervical Cerclage With Vaginal Progesterone in Asymptomatic Twin Pregnancies With a Sonographic Short Cervix
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, Principal Investigator, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: aswu/190/18
Record Dates: First submitted 2018-12-18; First posted 2018-12-20 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Twin; Pregnancy, Affecting Fetus or Newborn
Keywords: Preterm birth; Twin gestation; Vaginal progesterone; cervical cerclage
MeSH Terms: conditions — Premature Birth | interventions — Cerclage, Cervical

STUDY DESIGN:
Intervention Model Description: A randomized clinical trial
Masking Description: A randomized clinical trial open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cervical cerclage (Active Comparator): Cervical cerclage in twin pregnancy with transvaginal cervical length ≤25mm
  Interventions: Procedure: Cervical cerclage
- vaginal progesterone (Active Comparator): Daily vaginal progesterone 400mg from diagnosis of the short cervix to 36 weeks
  Interventions: Drug: vaginal progesterone
- Cervical cerclage plus vaginal progesterone (Active Comparator): Cervical cerclage in twin pregnancy with transvaginal cervical length ≤25mm plus Daily vaginal progesterone 400mg from diagnosis of the short cervix to 36 weeks
  Interventions: Procedure: Cervical cerclage; Drug: vaginal progesterone

INTERVENTIONS:
Procedure: Cervical cerclage — Cervical cerclage indicated by short cervix ≤25mm
  Other Names: Active Comparator
  Arms: Cervical cerclage; Cervical cerclage plus vaginal progesterone
Drug: vaginal progesterone — Daily vaginal progesterone 400mg from diagnosis of short cervix to 36 weeks
  Other Names: Active Comparator
  Arms: Cervical cerclage plus vaginal progesterone; vaginal progesterone

SUMMARY:
The objective of the present study is to evaluate the effectiveness of vaginal progesterone and cervical cerclage each alone and in combination in improving gestational age in twin pregnancy and its subsequent impact on perinatal outcome.

DETAILED DESCRIPTION:
There is a lack of effective, evidence-based interventions for the prevention of preterm birth in twin pregnancies. There is limited evidence for the use of vaginal progesterone and cervical cerclage, and the cervical pessary is currently only used within a research setting. There are no reported trials comparing the effectiveness of each of these interventions against each other, whether in isolation or in combination. Research is needed to further evaluate the benefit of the cervical pessary and the use of cervical cerclage in twins of women with a short cervix. A recent article by Stock et al.concludes by advising clinicians to share with women the uncertainty of methods to prevent PTB in multiple pregnancies, and offer the opportunity to participate in clinical trials. So the objective of the present study is to evaluate the effectiveness of vaginal progesterone and cervical cerclage each alone and in combination in improving gestational age in twin pregnancy and its subsequent impact on perinatal outcome.

ELIGIBILITY:
Inclusion Criteria:

* Women pregnant in dichorionic twins.
* Transvaginal sonographic cervical length is <25 mm at 16-20 weeks gestational age.
* No symptoms, signs or other risk factors for preterm labor

Exclusion Criteria:

* Age < 18 years or > 45 years.
* Known allergy or contraindication (relative or absolute) to progesterone therapy.
* Monochorionic twins.
* Known major fetal structural or chromosomal abnormality.
* Intrauterine death of one fetus or death of both fetuses.
* Fetal reduction in the current pregnancy.
* Medical conditions that may lead to preterm delivery.
* Rupture of membranes.
* Vaginal bleeding

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women pregnant in dichorionic twins
Enrollment: 300 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Preterm labor before 34 weeks | Up to 34 weeks gestational age
  Number of patients with preterm birth before 34 weeks gestations

SECONDARY OUTCOMES:
Neonatal respiratory distress syndrome | At birth
  number of neonatal respiratory distress syndrome
Early neonatal death | within one month postpartum
  number babies died in the neonatal period

CONTACTS AND LOCATIONS:
Overall Officials: hany f sallam, md, Principal Investigator — Aswan University Hospital
Locations (1):
- Aswan University, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: Undecided